CLINICAL TRIAL: NCT06523985
Title: The Feasibility of Using the National PulsePoint Cardiopulmonary Resuscitation Responder Network to Facilitate Overdose Education and Naloxone Distribution
Brief Title: The Feasibility of Using the PulsePoint to Facilitate Overdose Education and Naloxone Distribution
Acronym: PP-OD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jon Agley, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R34DA058162 (NIH); R34DA058162 (NIH)
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Carrying Naloxone/Narcan on Their Person or in Their Vehicle; Being Trained to Respond to an Opioid Overdose

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard layperson messaging (Arm 1) (Active Comparator): Users randomized to arm 1 will receive standard monthly recruitment push messages. These push messages will differ from the certification messages because they will contain language intended to foster engagement with OEND services (eg, to get trained and carry naloxone) alongside the link to a landing page.
  Interventions: Behavioral: Push messages (standard)
- Customized layperson messaging (Arm 2) (Experimental): Arm 2 will follow the same procedures that are described for arm 1 but will use separate messaging. Specifically, the push messages and landing page will contain additional, brief messages that specifically provide factual information that counteracts misperceptions about overdose and naloxone.
  Interventions: Behavioral: Push messages (customized)
- Control arm (Arm 3) (No Intervention): Arm 3 functions as the control arm and will not receive any monthly recruitment messaging or encouragement.

INTERVENTIONS:
Behavioral: Push messages (standard) — Push messages will be developed based on best practice recruitment principles in cooperation with an external marketing team and then reviewed and finalized by the study team. Messages will be different each month and sent across 12 months. The monthly time frame was selected based on our need to balance contact with responders and research or expert opinions on push messaging saturation.
  Arms: Standard layperson messaging (Arm 1)
Behavioral: Push messages (customized) — These messages are similar to content in the standard push messages but are customized to address common misperceptions about opioid overdose and naloxone.
  Arms: Customized layperson messaging (Arm 2)

SUMMARY:
This study is a feasibility trial to assess whether, in a random sample of 180 agencies where PulsePoint is already active, revised procedures (hereinafter PulsePoint-OD) to facilitate opioid overdose and naloxone distribution (OEND) can successfully recruit first responder agencies and layperson responders. For this study, agency refers to a single implementation site where PulsePoint is active and that is bound by the service area or jurisdiction of the first responder agency collaborating with PulsePoint.

The study will test the following hypotheses:

H1: more first responder agencies will be successfully recruited by arm 2 than by arm 1.

H2: more layperson responders will report engaging with OEND programming in arm 2 than in arms 1 or 3 and in arm 1 than in arm 3 [only this hypothesis is covered by the IRB, hypothesis 1 is not human subjects research].

DETAILED DESCRIPTION:
A full, detailed description of the study protocol and preregistered procedures is located in our formal protocol paper (https://doi.org/10.2196/57280) which is also cited at the end of this specific registration.

All specific language throughout this document is derived directly (verbatim) from the protocol paper, which is our controlling, planned preregistration document for this project.

ELIGIBILITY:
Layperson responders who are part of the PulsePoint system register with a local first responder agency using their smartphone. Anyone who is registered with a PulsePoint agency randomly selected for this project is included. Most layperson responders (eg, those who are not also off-duty first responders themselves) are only alerted to incidents in public spaces. No identifying information is collected from these users except the unique ID of the device.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Certification of receiving OEND programming and naloxone carrying | 12 months
  At baseline, we will calculate the ratio of persons certifying that they are trained (numeric count of N) compared to the total number of push message recipients (T), the ratio of persons certifying that they carry naloxone (numeric count of C) compared to the total number of push message recipients (T), and the ratio of individuals who clicked on the link (O) compared to the total number of push message recipients (T). Separately at 6- and 12-month follow-ups, the numbers of certifications of training and carrying naloxone (N and C, respectively) that were submitted compared to the numbers of push recipients (T) in each period (tracked by D) and the ratio of individuals who clicked on the link (O) each month compared to the number of total push message recipients (T). Our outcome variables are ratios: X = (N / T) for each value of D (0, 1, or 2) and Y = (C / T) for each value of D. The ratio Z = (O / T) is a covariate representing engagement with push messages at each value of D.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Agley, Principal Investigator — Indiana University
Locations (1):
- Indiana University Bloomington, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified raw data will be provided alongside publications using those data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available in perpetuity once published.
Access Criteria: Data will be fully anonymous (in ratio format) and access will not be curtailed.

REFERENCES:
- [Background] Agley J, Henderson C, Seo DC, Parker M, Golzarri-Arroyo L, Dickinson S, Tidd D. The Feasibility of Using the National PulsePoint Cardiopulmonary Resuscitation Responder Network to Facilitate Overdose Education and Naloxone Distribution: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Mar 29;13:e57280. doi: 10.2196/57280. PMID 38551636
- See also: Open Science Framework Preregistration — https://doi.org/10.17605/OSF.IO/EGN3Z